CLINICAL TRIAL: NCT02873104
Title: Pivotal Study of the truSculpt Radiofrequency Device for Circumferential Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-16-TS11
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2017-02

CONDITIONS: Abdominal Fat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment (Active Comparator): truSculpt rf device, therapeutic settings
  Interventions: Device: truSculpt rf device
- Sham (Sham Comparator): truSculpt rf device, non-therapeutic settings
  Interventions: Device: truSculpt rf device

INTERVENTIONS:
Device: truSculpt rf device — radiofrequency device

SUMMARY:
To evaluate the safety and efficacy of the Cutera truSculpt radiofrequency device for circumferential reduction.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate efficacy and safety of treatment with the Cutera truSculpt RF device for circumferential reduction in the abdominal and flank region.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 24 to 60 years of age (inclusive). Fitzpatrick Skin Type I - VI. Has visible fat bulges on the abdomen and palpable fat pockets superior to iliac crest located bilaterally in the lower back flank region Has a Body Mass Index (BMI) ≥ 20 and ≤ 30 Non-smoking for at least 6 months and willing to refrain from smoking for the duration of the study.

Subject must agree to not undergo any other procedure(s) in the abdominal and flank region during the study period.

Subject must be able to read, understand and sign the Informed Consent Form. Subject must adhere to the follow-up schedule and study instructions. Subject must adhere to the same diet and/or exercise routine throughout the study, and agree to maintain the same weight throughout the study, within 5% of baseline weight measurement.

Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.

Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant.

Exclusion Criteria:

* Participation in a clinical trial of another device or drug within 6 months of study participation, or during the study period.

Any type of prior cosmetic treatment to the target area within 12 months of study participation e.g., radiofrequency, cryolysis or light-based treatments.

Any prior invasive cosmetic surgery to the target area, such as liposuction. Currently taking medications or supplements for weight-loss or metabolism support/enhancement or has a history of taking such medications or supplements within 3 months.

Has a pacemaker, internal defibrillator, implantable cardioverter-defibrillator, nerve stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant.

Has metal implant(s) within the body, such as surgical clips, plates and screws, intrauterine device (IUD), artificial heart valves or artificial joints.

Significant concurrent illness, such as diabetes mellitus, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders.

Diagnosed or documented immune system disorders. History of any disease or condition that could impair wound healing. History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.

History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing.

Infection, dermatitis, rash or other skin abnormality in the target area. Currently undergoing systemic chemotherapy or radiation treatment for cancer, or history of treatment in the target area within 3 months of study participation.

Pregnant or currently breastfeeding. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 24 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cutera Research Center, Brisbane, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Sham
Started | 47 | 23
Completed | 46 | 23
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Sham | Total
Number analyzed (Participants) | 47 | 23 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 23 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 8 | 45
  Male | 10 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Difference in Circumferential Measurement Related to Sham and Therapeutic Group at 12 Weeks Post-treatment
Description: Change in Abdominal Circumferential Measurement Related to Sham and Therapeutic Group at 12 Weeks Post-treatment minus Baseline Measurement
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: cm
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 46 | 23
cm | 1.9 (0.1) | 0 (0.1)

2. Secondary Outcome: Subject Assessment of Improvement for Both Sham Group and Therapeutic Group at 12 Weeks Post-treatment.
Description: Comparison of the average subject improvement score for the sham group and the therapeutic group at 12 weeks post-treatment using a 0 - 4 improvement scale where 0 equals "no change" and 4 equals "Very Significant Improvement".
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 46 | 23
units on a scale | 2.4 (1) | 1 (1.5)

3. Secondary Outcome: Subject Satisfaction Level for Both Sham Group and Therapeutic Group at 12 Weeks Post-treatment.
Description: Comparison of the average subject satisfaction level for the sham group and therapeutic group at 12 weeks post-treatment, using a 1 - 5 scale where 1 equals "very dissatisfied" and 5 equals "very satisfied".
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 46 | 23
units on a scale | 4.1 (0.8) | 3.3 (0.9)

4. Secondary Outcome: Subject Discomfort and Pain Levels During Treatment
Description: Comparison of the average pain levels during treatment for the sham group and therapeutic group at 12 weeks post-treatment, using a 0 - 10 scale where 0 equals "No pain" and 10 equals "Worst possible pain".
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 47 | 23
units on a scale | 5.75 (0.9) | 1.1 (0.3)

ADVERSE EVENTS:
Arm/Group | Treatment | Sham
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/23
Other Adverse Events (participants affected / at risk) | 47/47 | 23/23
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=47) | Sham (N=23)
Erythema (Skin and subcutaneous tissue disorders) | 47 (47) | 23 (23)
Edema (Skin and subcutaneous tissue disorders) | 47 (47) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes